CLINICAL TRIAL: NCT06783244
Title: Low Versus Standard Intraabdominal Pressure in Robot-assisted Colorectal Cancer Surgery: A Double Blinded Randomized Clinical Trial
Brief Title: Low Versus Standard Intraabdominal Pressure in Robot-assisted Colorectal Cancer Surgery
Acronym: LIPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Victoria Rosberg (Other)
Responsible Party: Sponsor-Investigator, Victoria Rosberg, Medical Doctor and PhD student, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: H-24073961
Record Dates: First submitted 2024-12-20; First posted 2025-01-20 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; robot-assisted surgery; intraabdominal pressure
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low pressure (8 mmHg) (Active Comparator): Patients diagnosed with colorectal cancer undergoing robot-assisted surgery performed with low intraabdominal pressure (8 mmHg)
  Interventions: Other: Low intraabdominal pressure (8 mmHg)
- Standard pressure (12 mmHg) (No Intervention): Patients diagnosed with colorectal cancer undergoing robot-assisted surgery performed with standard intraabdominal pressure (12 mmHg)

INTERVENTIONS:
Other: Low intraabdominal pressure (8 mmHg) — Only difference in treatment is the lower level of intraabdominal pressure by which the procedure is performed. The intervention does not change the treatment. The surgical procedure is performed due to Danish national guidelines and remains the same in the two arms.
  Arms: Low pressure (8 mmHg)

SUMMARY:
The goal of this clinical trial is to investigate the influence of low intraabdominal pressure (compared to standard intraabdominal pressure) during robot-assisted colorectal cancer surgery on patients wellbeing after surgery. Patients included are diagnosed with colon- or rectal cancer, and scheduled for curatively intended surgery. The main question the trial aims to answer is:

Does low intraabdominal pressure during robot-assisted colorectal cancer surgery increase the patients wellbeing after surgery?

Researchers will compare low intraabdominal pressure (8 mmHg) to standard intraabdominal pressure (12 mmHg) to see if there is a difference in quality of recovery scores, pain scores and analgetic consumption.

Participants will be asked to fill out the Quality of Recovery 15 (QoR15) questionnaire 8 hours, 24 hours and 48 hours after surgery. Furthermore, patients will be asked to evaluate abdominal pain and shoulder tip pain using the visual analog scale (VAS).

DETAILED DESCRIPTION:
1. Introduction

   Colorectal cancer is the third most frequent malignancy worldwide with an increasing incidence. Surgical resection is considered the gold standard for the cure of colorectal cancer. It is well recognized that an uneventful postoperative course is pivotal for a favorable prognosis. The length of stay (LOS) after colorectal cancer surgery has traditionally been between 1 and 2 weeks after surgery. This period has rightfully received considerable attention, and in the 2000s, Enhanced Recovery after Surgery (ERAS) protocols emerged as evidence-based perioperative practice guidelines designed to optimize the postoperative outcome and thereby shorten LOS. The ERAS principle is based on multimodal strategies, which collectively accelerates recovery and helps patients return to their baseline physical function more rapidly. ERAS has significantly reduced LOS without compromising patient safety or satisfaction. Minimally invasive surgery (MIS), including laparoscopic and robot-assisted techniques, is now an integral part of modern ERAS and a cornerstone of colorectal cancer surgery.

   In general, MIS has been proven to reduce morbidity, postoperative pain and analgesic consumption, duration of hospital stay and patient satisfaction after colectomy. To ensure proper visceral exposure during minimal invasive surgery CO2 needs to be insufflated into the abdominal cavity. However, the insufflation and the inevitable increased intraabdominal pressure has been associated with postoperative shoulder pain and deep abdominal pain. The standard level of intraabdominal pressure is set around 12 mmHg in most situations and lowering the pressure could possibly decrease the morbidity associated with insufflation.

   The first studies investigating the benefits and disadvantages of low-pressure laparoscopic surgery were performed in patients undergoing cholecystectomy and three major meta-analyses have suggested advantages in low-pressure surgery including reduced postoperative pain, analgesic use, and a slight reduction in length of stay.

   There are only few studies on low pressure colorectal surgery and even fewer using the robotic platform, where the increased dexterity improves the surgical conditions in smaller confined spaces, which may be the result of lowering the pressure. Previously, Diaz-Cambronero et al. demonstrated that 78% of these procedures could safely be completed at 8 mmHg.

   In 2021, S. Celarier and colleagues published The PAROS trial, which was the first prospective randomized trial on low (7 mmHg) versus standard (12 mmHg) intraabdominal pressure in laparoscopic colorectal surgery. The length of stay was significantly decreased in the low-pressure group along with postoperative pain and analgesic consumption. They argued that low pressure should become standard of care in laparoscopic colectomy. Furthermore, low intraabdominal pressure did not compromise peri- or postoperative outcomes, operating time, or oncological safety. A year later, the RECOVER study, a randomized controlled trial, re-ported a clear advantage of low (8 mmHg) intraabdominal pressure in combination with deep neuromuscular blockage during laparoscopic colorectal surgery. This combination proved to be safe and improve the postoperative patient-reported quality of recovery.

   A recent systematic review and meta-analysis found no superiority of low- compared with standard/high pressure during laparoscopic colorectal cancer surgery on LOS, however, postoperative pain and analgesic consumption were not investigated.

   Current recommendation is to use the lowest possible intraabdominal pressure allowing suffi-cient exposure of the operative field, rather than using a routine pressure. This recommendation was published more than 20 years ago, however, in the 2018 ERAS Society guideline for Perioperative Care in Elective Colorectal Surgery it was stated that evidence for reducing intraabdominal pressure is low.

   The used standard pressure of 12 mmHg may be higher than necessary, leaving a potential to reduce pressure and thereby facilitate faster recovery with decreased postoperative pain and increased physical well-being at the time of discharge.
2. Objective and perspective

   The objective of the present study is to investigate the role of low intraabdominal pressure during robot-assisted colorectal cancer surgery on immediate postoperative recovery.

   By challenging the practice of using a standard pressure of 12 mmHg, this trial has the potential to optimize postoperative care and patient satisfaction in robot-assisted colorectal cancer surgery, paving the way for advancements beyond ERAS, potentially enabling same day surgery for selected patients with colorectal cancer.
3. Early patient involvement

   Before initiating the trial, a group of surviving patients previously treated for colorectal cancer at our institution, will be invited to take part in a group interview, with the purpose of giving their important view on the selection of the study endpoints including the rationale for the primary endpoint and possible missed endpoints important for the patients.

   This group of patients will be identified in our local cancer database. An equal gender balance will be ensured, younger and elder patients will be represented, and it will furthermore be ensured that both right and left/rectum resection is represented.

   After the study data have been concluded and the data have been analyzed according to the agreed plan, the same group of patients will be invited to participate in a group presentation of the study results and with the opportunity to give their view on how the results should be interpreted.
4. Experimental plan

4.1. Study design

Investigators aim to conduct a multicenter, double blinded, prospective, randomized trial including patients undergoing robotic colorectal cancer resection, involving collaborating departments from Sweden, Norway and Denmark.

Patients scheduled for elective robot assisted colon or rectal cancer resection will be assessed for eligibility and if inclusion criteria are met patients are included after informed consent. Participants will by randomization be included in a low-pressure group (8 mmHg) or a standard pressure group (12 mmHg) and participant will be stratified according to location of the tumor, right or left/rectal.

It is important to underline, that participants included will receive same standardized surgical treatment as if not included. The operational strategy and procedure will be performed due to national guidelines by a certified colorectal cancer surgeon.

4.5 Data collection and storage

A dedicated REDCap database will be created for online registration using an electronic case report form (eCRF). The case report form will obtain data in regard to in- and exclusion criteria, primary and secondary endpoints and general health, i.e. co-morbidities and data regard-ing the specific case peri and post operation.

Only after informed and written consent, data will be collected directly to the database by clinicians involved in the surgical procedure, who thereby have access to the journal. Beyond this, only the applicant, Victoria Rosberg (VR), and supervisor Peter-Martin Krarup (PMK) are authorized to directly access the patient's journal (including electronical journal) for the purpose of retrieving data necessary for the project. VR and PMK are the only individuals with access to any records registered (i.e. CPR numbers) in the database and will therefore be the sole persons authorized to access patient journals after end procedure or discharge in order to retrieve any missing data. Investigators expect to access 200 medical journals in total (see under power calculation).

4.6 Requirements of participating departments

In this study, investigators aim to standardize the perioperative course therefore, participating surgeons should be experts in robotic colorectal surgery and study operations should not be used for training. For insufflation, the AirSeal system (Conmed) should be used to ensure a staple and uniform intraabdominal pressure and minimize differences between centers.

Participating centers should adhere to the latest ERAS protocol including urinary catheter re-moval immediately after surgery, early mobilization, and nutrition (day 0).

4.7 Patient consent, randomization and blinding

The staff and research personnel receive the protocol to identify patients eligible for inclusion. Inclusion of participants is initiated during the pre-operation appointment. The surgeon informs eligible participants regarding the intervention, the purpose of the study and the foreseeable risks and hypothesized benefits. Participants will have the opportunity to get any question an-swered and are free to be accompanied by relatives if wished.

If a patient consent to participation, a signed informed consent will be obtained and kept in an area inaccessible to third parties. Participants will be given a copy of the informed consent and may at all times withdraw their consent. Participants who decide to withdraw their con-sent will still receive the surgical treatment they were planned to undergo, however, without intervention and data will not be collected to the database.

On the day of surgery, the operating nurse will register the patient in the RED Cap database prior to the procedure, and the database will subsequently assign the patient to a randomiza-tion group. Randomization will thereby be performed using a computer-generated randomiza-tion within the Red Cap database, accessible from the operating room. The operating nurse oversees the randomization. After first insufflation and port placement at 12 mmHg, CO2 is exsufflated and randomization is commenced. The view to the pressure monitor blocked for the surgeons by the operating nurse. The nurse changes the pressure according to randomi-zation, standard (12 mmHg) or low (8 mmHg). The operating nurse will, at all times, be able to view the current intraabdominal pressure.

During the operation, the surgeon is at all times allowed to raise the pressure to 12 mmHg if exposure is poor and operational safety is compromised. For participants in the standard pressure group, the nurse will simulate a change in pressure. Blinding is kept. The surgeon can at all time unblind the patient if necessary.

4.8 Power calculation

To detect a clinically significant between-group difference of 10% in the primary endpoint, QoR15, the required sample size was calculated on the following parameters; a mean value in QoR15 of 97, measured six hours postoperatively in a previous study, a standard deviation in outcome of 23 between baseline- and eight hours postoperatively, a power of 80%, and a type I error of 5%. Based on above parameters, 84 participants in each arm (low- versus standard pressure) is required. To account for dropouts, the number of participants is in-creased to 200 (100 in each arm). No interim analysis is planned.

5 Ethical considerations

The study will not commence before approval from the Committee of Health Research Ethics. All participants will need to sign informed consent and can at any time withdraw their consent. All patient data will be processed and stored in accordance with the General Data Protection Regulation (GDPR). Any patient data handled outside of either the encrypted remote-access registry data server or the RED Cap study database will be fully anonymized and han-dled according to appropriate regulations.

5.1 Patient risk assessment

The intervention has previously demonstrated safety in laparoscopic procedures (see introduction). Therefore, it is considered to pose minimal risk to the patient. Furthermore, the intervention is easily reversible, and the surgeon retains the ability to adjust the pressure at any time during the surgery, should it be deemed necessary to ensure safety and maintain operational quality.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* a diagnosis of colorectal cancer
* scheduled for curative intended robot-assisted resection

Exclusion Criteria:

* BMI above 35
* inability to fulfill QoR15 questionnaire
* construction of a stoma either proactive or permanent
* metastatic cancer disease
* recieving neoadjuvant treatment
* previous multiple abdominal operations defined as 3 or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery 15 (QoR15) questionnaire 8 hours after surgery | From end of surgery until 8 hours later
  The quality of recovery 15 (QoR15) questionnaire is a composite patient-centered rating scale measuring different important aspects of the postoperative recovery and fulfils the require-ments for outcome measurement instruments in clinical trials. The questionnaire consist of 15 questions, each being answered on a scale from 0-10. Thereby summed scores ranges from 0 to 150; 0 being the worst outcome and 150 being the best outcome. The questionnaire has been translated and validated in a Danish version and preserved the same validity, reliability, and high degree of responsiveness and clinical feasibility.

SECONDARY OUTCOMES:
QoR15 questionnaire 24 og 48 hours after surgery | From end of surgery until 24 and 48 hours later
  The quality of recovery 15 (QoR15) questionnaire is a composite patient-centered rating scale measuring different important aspects of the postoperative recovery and fulfils the require-ments for outcome measurement instruments in clinical trials. The questionnaire consist of 15 questions, each being answered on a scale from 0-10. Thereby summed scores ranges from 0 to 150; 0 being the worst outcome and 150 being the best outcome. The questionnaire has been translated and validated in a Danish version and preserved the same validity, reliability, and high degree of responsiveness and clinical feasibility.
Postoperative pain score | From end of surgery until at 8 hours, 24 hours and 48 hours after surgery
  Postoperative pain scores measured using the visual analog scale (VAS). VAS ranges from 0 to 10, where 0 is no pain and 10 is the worst possible pain.
Postoperative opioid consumption | End of surgery until 3 days after surgery. Assessed up to 6 months after surgery.
  Data on type and amount of opiod consumption after surgery.
Change in intraabdominal pressure during surgery | From operation start until end of surgery. Assessed up to 6 months after surgery.
  If the surgeon askes for the pressure to be changed during surgery this will be recorded.
Operation time | From operation start until end of surgery. Assessed up to 6 months after surgery.
  Duration time of the procedure performed
Surgeons experience | Assessed immediately after surgery
  The surgeon fulfills a short questionnaire (approximately 5 questions) on his/her subjective evaluation of how the procedure went. Answers are given as yes or no. No scores are given.
Postoperative complications | End of surgery until discharge. Assessed up to 6 months after surgery.
  Postoperative complications will be measured using the Clavien Dindo score.
Intensive care unit stays | Until 30 days after surgery. Assessed up to 6 months after surgery.
  If the patient is admitted to an intensive care unit within 30 days after surgery this will be recorded
30-day mortality rate | Until 30 days after surgery. Assessed up to 6 months after surgery.
  If a patient dies within 30 days after surgery this will be recorded
Length of stay (LOS) | From admission until discharge. Assessed up to 6 months after surgery.
  The number of days the patient is admitted to the hospital in relation to the surgery
EQ-5D-5L questionnaire | Upon discharge from hospital. Assessed up to 6 months after surgey.
  The Euro Quality of Life 5 Dimension 5 Level (EQ-5D-5L) is a self-reported, health related survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each domain there is 5 possible answers (5 levels): no problems, slight problems, moderate problems, severe problems and extreme problems The patient will be asked to fill out the questionnaire when he/she is discharged from the hospital.
30-day readmission rates | Until 30 days after surgery. Assessed up to 6 months after surgery.
  If patients are readmitted to the hospital within 30 days after surgery this will be recorded
Patient satisfaction assessment | From end of surgery until participant is discharged. Assessed up to 6 months after surgery.
  At discharge patients will be asked if they are overall satisfied with the treatment (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Disease Center, Copenhagen University Hospital, Bispebjerg, Copenhagen NV, Denmark

REFERENCES:
- [Background] Dohrn N, Yikilmaz H, Laursen M, Khesrawi F, Clausen FB, Sorensen F, Jakobsen HL, Brisling S, Lykke J, Eriksen JR, Klein MF, Gogenur I. Intracorporeal Versus Extracorporeal Anastomosis in Robotic Right Colectomy: A Multicenter, Triple-blind, Randomized Clinical Trial. Ann Surg. 2022 Nov 1;276(5):e294-e301. doi: 10.1097/SLA.0000000000005254. Epub 2021 Oct 13. PMID 35129520
- [Background] Kleif J, Edwards HM, Sort R, Vilandt J, Gogenur I. Translation and validation of the Danish version of the postoperative quality of recovery score QoR-15. Acta Anaesthesiol Scand. 2015 Aug;59(7):912-20. doi: 10.1111/aas.12525. Epub 2015 Apr 13. PMID 25867135
- [Background] Kleif J, Waage J, Christensen KB, Gogenur I. Systematic review of the QoR-15 score, a patient- reported outcome measure measuring quality of recovery after surgery and anaesthesia. Br J Anaesth. 2018 Jan;120(1):28-36. doi: 10.1016/j.bja.2017.11.013. Epub 2017 Nov 22. PMID 29397134
- [Background] Neudecker J, Sauerland S, Neugebauer E, Bergamaschi R, Bonjer HJ, Cuschieri A, Fuchs KH, Jacobi Ch, Jansen FW, Koivusalo AM, Lacy A, McMahon MJ, Millat B, Schwenk W. The European Association for Endoscopic Surgery clinical practice guideline on the pneumoperitoneum for laparoscopic surgery. Surg Endosc. 2002 Jul;16(7):1121-43. doi: 10.1007/s00464-001-9166-7. Epub 2001 May 20. PMID 12015619
- [Background] Hamid M, Mostafa OES, Mohamedahmed AYY, Zaman S, Kumar P, Waterland P, Akingboye A. Comparison of low versus high (standard) intraabdominal pressure during laparoscopic colorectal surgery: systematic review and meta-analysis. Int J Colorectal Dis. 2024 Jul 10;39(1):104. doi: 10.1007/s00384-024-04679-8. PMID 38985344
- [Background] Albers KI, Polat F, Helder L, Panhuizen IF, Snoeck MMJ, Polle SBW, de Vries H, Dias EM, Slooter GD, de Boer HD, Diaz-Cambronero O, Mazzinari G, Scheffer GJ, Keijzer C, Warle MC; RECOVER Study Collaborators. Quality of Recovery and Innate Immune Homeostasis in Patients Undergoing Low-pressure Versus Standard-pressure Pneumoperitoneum During Laparoscopic Colorectal Surgery (RECOVER): A Randomized Controlled Trial. Ann Surg. 2022 Dec 1;276(6):e664-e673. doi: 10.1097/SLA.0000000000005491. Epub 2022 Jul 13. PMID 35822730
- [Background] Celarier S, Monziols S, Celerier B, Assenat V, Carles P, Napolitano G, Laclau-Lacrouts M, Rullier E, Ouattara A, Denost Q. Low-pressure versus standard pressure laparoscopic colorectal surgery (PAROS trial): a phase III randomized controlled trial. Br J Surg. 2021 Aug 19;108(8):998-1005. doi: 10.1093/bjs/znab069. PMID 33755088
- [Background] Diaz-Cambronero O, Flor Lorente B, Mazzinari G, Vila Montanes M, Garcia Gregorio N, Robles Hernandez D, Olmedilla Arnal LE, Argente Navarro MP, Schultz MJ, Errando CL; IPPColLapSe study group. A multifaceted individualized pneumoperitoneum strategy for laparoscopic colorectal surgery: a multicenter observational feasibility study. Surg Endosc. 2019 Jan;33(1):252-260. doi: 10.1007/s00464-018-6305-y. Epub 2018 Jun 27. PMID 29951750
- [Background] Gurusamy KS, Vaughan J, Davidson BR. Low pressure versus standard pressure pneumoperitoneum in laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2014 Mar 18;2014(3):CD006930. doi: 10.1002/14651858.CD006930.pub3. PMID 24639018
- [Background] Ozdemir-van Brunschot DM, van Laarhoven KC, Scheffer GJ, Pouwels S, Wever KE, Warle MC. What is the evidence for the use of low-pressure pneumoperitoneum? A systematic review. Surg Endosc. 2016 May;30(5):2049-65. doi: 10.1007/s00464-015-4454-9. Epub 2015 Aug 15. PMID 26275545
- [Background] Hua J, Gong J, Yao L, Zhou B, Song Z. Low-pressure versus standard-pressure pneumoperitoneum for laparoscopic cholecystectomy: a systematic review and meta-analysis. Am J Surg. 2014 Jul;208(1):143-50. doi: 10.1016/j.amjsurg.2013.09.027. Epub 2014 Jan 16. PMID 24503370
- [Background] Ergun M, Berkers AW, van der Jagt MF, Langenhuijsen JF, van Ozdemir-Brunschot D, van der Vliet JA, D'Ancona FC, Warle MC. Components of pain assessment after laparoscopic donor nephrectomy. Acta Anaesthesiol Scand. 2014 Feb;58(2):219-22. doi: 10.1111/aas.12236. Epub 2013 Dec 6. PMID 24308727
- [Background] Bisgaard T, Klarskov B, Rosenberg J, Kehlet H. Characteristics and prediction of early pain after laparoscopic cholecystectomy. Pain. 2001 Feb 15;90(3):261-269. doi: 10.1016/S0304-3959(00)00406-1. PMID 11207398
- [Background] Lacy AM, Garcia-Valdecasas JC, Delgado S, Castells A, Taura P, Pique JM, Visa J. Laparoscopy-assisted colectomy versus open colectomy for treatment of non-metastatic colon cancer: a randomised trial. Lancet. 2002 Jun 29;359(9325):2224-9. doi: 10.1016/S0140-6736(02)09290-5. PMID 12103285
- [Background] Klarenbeek BR, Veenhof AA, Bergamaschi R, van der Peet DL, van den Broek WT, de Lange ES, Bemelman WA, Heres P, Lacy AM, Engel AF, Cuesta MA. Laparoscopic sigmoid resection for diverticulitis decreases major morbidity rates: a randomized control trial: short-term results of the Sigma Trial. Ann Surg. 2009 Jan;249(1):39-44. doi: 10.1097/SLA.0b013e31818e416a. PMID 19106674
- [Background] Veldkamp R, Kuhry E, Hop WC, Jeekel J, Kazemier G, Bonjer HJ, Haglind E, Pahlman L, Cuesta MA, Msika S, Morino M, Lacy AM; COlon cancer Laparoscopic or Open Resection Study Group (COLOR). Laparoscopic surgery versus open surgery for colon cancer: short-term outcomes of a randomised trial. Lancet Oncol. 2005 Jul;6(7):477-84. doi: 10.1016/S1470-2045(05)70221-7. PMID 15992696
- [Background] Kang SB, Park JW, Jeong SY, Nam BH, Choi HS, Kim DW, Lim SB, Lee TG, Kim DY, Kim JS, Chang HJ, Lee HS, Kim SY, Jung KH, Hong YS, Kim JH, Sohn DK, Kim DH, Oh JH. Open versus laparoscopic surgery for mid or low rectal cancer after neoadjuvant chemoradiotherapy (COREAN trial): short-term outcomes of an open-label randomised controlled trial. Lancet Oncol. 2010 Jul;11(7):637-45. doi: 10.1016/S1470-2045(10)70131-5. Epub 2010 Jun 16. PMID 20610322
- [Background] Panis Y, Maggiori L, Caranhac G, Bretagnol F, Vicaut E. Mortality after colorectal cancer surgery: a French survey of more than 84,000 patients. Ann Surg. 2011 Nov;254(5):738-43; discussion 743-4. doi: 10.1097/SLA.0b013e31823604ac. PMID 21997816
- [Background] Adamina M, Kehlet H, Tomlinson GA, Senagore AJ, Delaney CP. Enhanced recovery pathways optimize health outcomes and resource utilization: a meta-analysis of randomized controlled trials in colorectal surgery. Surgery. 2011 Jun;149(6):830-40. doi: 10.1016/j.surg.2010.11.003. Epub 2011 Jan 14. PMID 21236454
- [Background] Lv L, Shao YF, Zhou YB. The enhanced recovery after surgery (ERAS) pathway for patients undergoing colorectal surgery: an update of meta-analysis of randomized controlled trials. Int J Colorectal Dis. 2012 Dec;27(12):1549-54. doi: 10.1007/s00384-012-1577-5. Epub 2012 Sep 22. PMID 23001161
- [Background] Zhuang CL, Ye XZ, Zhang XD, Chen BC, Yu Z. Enhanced recovery after surgery programs versus traditional care for colorectal surgery: a meta-analysis of randomized controlled trials. Dis Colon Rectum. 2013 May;56(5):667-78. doi: 10.1097/DCR.0b013e3182812842. PMID 23575408
- [Background] Basse L, Hjort Jakobsen D, Billesbolle P, Werner M, Kehlet H. A clinical pathway to accelerate recovery after colonic resection. Ann Surg. 2000 Jul;232(1):51-7. doi: 10.1097/00000658-200007000-00008. PMID 10862195
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Schoetz DJ Jr, Bockler M, Rosenblatt MS, Malhotra S, Roberts PL, Murray JJ, Coller JA, Rusin LC. "Ideal" length of stay after colectomy: whose ideal? Dis Colon Rectum. 1997 Jul;40(7):806-10. doi: 10.1007/BF02055437. PMID 9221857
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338